CLINICAL TRIAL: NCT06761573
Title: Bilateral Bispectral Index and Asymmetries in High Risk Patients for Posteoperative Delirium: An Observational, Prospective, Exploratory Study
Brief Title: Bilateral Bispectral Index, Asymmetries and Post-operative Delirium
Acronym: DELBIS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DELBIS
Record Dates: First submitted 2021-03-23; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction
Keywords: Bilateral Bispectral Index; Head&Neck Surgery; Plastic Surgery; Postoperative Delirium; Postoperative Cognitive Dysfunction; Interhemispheric asymmetries
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Complementary Therapies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patiets, undergoing head and neck surgery or plastic surgery, with high risk of POD: Each recruited patient, once on the operating bed, will be monitored with two BIS sensor, applied on the forehead in a non-invasive way, each for hemisphere.
  BIS Vista® monitor will be connected to our off-line laptop and software VitalDB will record: right&left BIS, BSR, Total Power, SEF, EMG, SQI and two BIS curves. Values of the study variables will be extract in these specific moments:(t1) BIS probe application (t2) 60" before GA administration (t3) 60" after myoresolution (t4) intubation (t5) surgical incision (t6) end of ipnosis (t7) 10 minutes after extubation.
  A daily follow-up for the first 5 post-operative days will verify the onset of POD and a telephone follow-up will be performed at 30 and 90 post-operative days to verify the onset of POD and POCD (CAM scale, 6-CIT scale and EQ50 for tracheostomized patients).
  Interventions: Device: Bilateral Bispetral Index Monitor will be applied on forehead of our patients, before surgery begins

INTERVENTIONS:
Device: Bilateral Bispetral Index Monitor will be applied on forehead of our patients, before surgery begins — In patients undergoing surgery and general anesthesia, the investigators want to examine -using bilateral BIS monitor- synthetic electroencephalographic differences between the two cerebral hemispheres (ASYM) to evaluate any correlation with the development of POD and POCD in the post-operative period.
  Other Names: CAM and CIT scales for diagnosis of POD and POCD will be post operativelly administrated to our patients

SUMMARY:
The primary objective of the study is to describe the value of interhemispheric asymmetry (ASYM), during the different intra- and peri-operative phases, in those patients who develop or do not develop post-operative delirium (POD) during the first 30 post-operative days and postoperative cognitive disfunction (POCD) in the first 90 post-operative days, in a population undergoing head&neck and plastic surgery with a priori increased probability of POD.

DETAILED DESCRIPTION:
Values of the study variables will be extract in these specific moments (considering a delay of thirty seconds between the in vivo phenomenon and the instrument): (t1) BIS probe application (t2) 60" before GA administration (t3) 60" after myoresolution (t4) intubation (t5) surgical incision (t6) end of ipnosis (t7) 10 minutes after extubation. Daily follow-up for the first five post-operative days is performed in order to verify the onset of POD and a telephone follow-up at thirty and ninety post-operative days in order to verify the onset of POD / POCD.

CAM scale will be used for the diagnosis of POD; while for the diagnosis of POCD, 6-CIT test will be used, the EQ50 test in the case of tracheostomized patients.

ELIGIBILITY:
Inclusion Criteria:

-Patients, undergoing head&neck surgery, who have at least 3 of the following criteria (to establish "a priori" increased risk of POD):

* Age> 70;
* Male sex; or ASA III;
* Smoker;
* High blood pressure;

Exclusion Criteria:

* ASA IV, V or ASA IE, IIE, IIIE (patients with anesthetic risk ASA>III and those undergoing urgent-emergency surgery will be excluded from the study);
* Past positive medical history for:

  * Stroke;
  * Dementia;
  * Cerebral aneurysm;
  * Intracranial mass;
  * Head trauma;
  * Epilepsy;
  * Diabetes mellitus;
  * Previous neurosurgical intervention;
  * Psychiatric illnesses requiring chronic treatment;
* Patients undergoing surgery in the previous two weeks;
* Patients whose hospitalization duration is estimated to be less than five days;
* Lack of understanding of the Italian language or English;
* Age <18 years.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll all patients undergoing head&neck surgery and plastic surgery, who meet the inclusion criteria. Patients will be screened and definitively enrolled after checking the inclusion and exclusion criteria. The study population, therefore, is represented by a minority of patients undergoing head&neck and plastic surgery, who have "a priori" increased risk of developing POD.
  The setting of the proposed study is the operating theaters of the operating block where the Anesthesia and Pain Therapy service is located, directed by Prof. Rita Maria Melotti, in pavilion 5 in the Policlinico Sant'Orsola-Malpighi in Bologna, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between ASYM (EEG-derived cerebral hemispheric asymmetries) at specific intraoperative timepoints and development of Postoperative Delirium (POD) or Postoperative Cognitive Dysfunction (POCD) | between 30 and 90 postoperative days
  Primary aim of the study is to describe values of ASYM, during different intraoperative phases, in patients who develop -or do not- POD within 5 postoperative days and POCD at 30 and 90 postoperative days. Bilateral BIS monitor records values of right and left BIS scores (dimensionless number EEG-derived from 0 to 100), therefore, the asymmetry between the two (ASYM) evaluated as the total power difference for the frequencies between 0 and 30 Hz between right and left hemisphere [Formula 1]. An asymmetry of 50% indicates the same power in both hemispheres; while an ASYM lower than 50% indicates a lower power in the left hemisphere than in the right.
  Formula 1:
  ASYM= total power left/(total power left+total power right) x 100 Dispersion of ASYM will be expressed as the mean right to left difference ±2 standard deviation.The statistical difference of the model will be evaluated with the use of ANOVA tests.

SECONDARY OUTCOMES:
Incidence of Postoperative Delirium (POD) and Postoperative Cognitive Dysfunction (POCD) in head&neck and plastic surgery | follow-up at 5, 30 and 90 postoperative days
  Secondary outcome of the study is to describe the incidence of Postoperative Delirium (POD) and Postoperative Cognitive Dysfunction (POCD) in patients undergoing head&neck and plastic surgery considered at "priori" high risk for development of POD with CAM scale and CIT-6 scale
Correlation between values of bilateral BSR, bilateral sBIS, bilateral sEMG at specific intraoperative timepoints and development of POD or POCD | Intraoperative phase: (t1) BIS probe application (t2) 60 seconds before GA administration (t3) 60 seconds after myoresolution (t4) intubation (t5) surgical incision (t6) end of ipnosis (t7) 10 minutes after extubation
  Secondary outcome is to evaluate differences in BIS monitor derived values: bilateral bilateral burst suppression ratio (BSR), bilateral bispectral index (BIS), bilateral elecromyography (sEMG), during the different intraoperative phases (repeated measures), between the group of patients who develop at least one episode of POD within 5 days and the group of patients who develop at least one episode of POCD within 90 postoperative days.
  Mean Differences ±2 standard deviation of these values will be evaluated in relation to the primary outcome (DPO and DCPO) through the use of a linear mixed effects model based on both inter-patient and inter-evaluation variability. The statistical difference of the model will be evaluated with the use of ANOVA tests.
Secondar outcomes is to evaluate inter and intra-patient variability of EEG-derived values at specific intraoperative timepoints | Intraoperative phase: (t1) BIS probe application (t2) 60 seconds before GA administration (t3) 60 seconds after myoresolution (t4) intubation (t5) surgical incision (t6) end of ipnosis (t7) 10 minutes after extubation
  Describe the inter- and intra-patient variability of the electroencephalographic derived values, during different intraoperative phases of general anesthesia.
  Differences in ASYM, bilateral BSR, bilateral sBIS, bilateral sEMG values during different peri-operative stages will be described (exploratory outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Paola Lauretta, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soehle M, Dittmann A, Ellerkmann RK, Baumgarten G, Putensen C, Guenther U. Intraoperative burst suppression is associated with postoperative delirium following cardiac surgery: a prospective, observational study. BMC Anesthesiol. 2015 Apr 28;15:61. doi: 10.1186/s12871-015-0051-7. PMID 25928189
- See also: PubMed — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4419445/